CLINICAL TRIAL: NCT00716911
Title: CMV Specific Cellular Immunity in Recipients of Allogeneic Bone Marrow Transplantation: Association of CMV-Specific HLA-Peptide Tetramer Binding With Cytotoxic T-Cell Function, CMV Infection and Other Clinical Events
Brief Title: Measuring Changes in Blood in Patients at High Risk of Cytomegalovirus Infection After Undergoing Donor Bone Marrow Transplant or Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: John A. Zaia, City of Hope Comprehensive Cancer Center
Purpose: Supportive Care
Other Study IDs: 99061; R01AI058148 (NIH); P30CA033572 (NIH); CHNMC-99061; CDR0000600022 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Nonneoplastic Condition
Keywords: cytomegalovirus infection; accelerated phase chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; splenic marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; stage I multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Cytomegalovirus Infections; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis | interventions — Ganciclovir; Polymerase Chain Reaction; Flow Cytometry; Immunologic Techniques; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ganciclovir
Genetic: polymerase chain reaction
Other: flow cytometry
Other: immunologic technique
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: assessment of therapy complications
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Tests that measure certain changes in blood in patients at high risk of cytomegalovirus infection may help doctors learn more about predicting cytomegalovirus infection after donor stem cell transplant.

PURPOSE: This clinical trial is studying tests that measure changes in the blood in patients at high risk of cytomegalovirus infection after undergoing donor bone marrow transplant or peripheral stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To document the quantitative characteristics of a cytomegalovirus (CMV)-specific HLA-peptide tetramer-binding assay (TBA) for cytotoxic T lymphocytes (CTLs) in patients who have undergone allogeneic bone marrow transplantation (BMT) or peripheral blood stem cell transplantation (PBSCT).
* To confirm the optimal TBA conditions for CTL characterization in these patients.
* To compare the TBA results for these patients with conventional assays for CTL functions.
* To compare CMV-specific TBA during the first 3 months after allogeneic BMT or PBSCT and to determine whether this binding function, in either donor or recipient, is a surrogate marker for protection from risk of CMV infection in these patients.
* To determine whether acquisition of CMV-specific TBA protects from risk for CMV disease in patients having active CMV infection after allogeneic BMT or PBSCT.

OUTLINE: This is a multicenter study. Patients accrue initially to cohort 1 until a sufficient number of stem cell transplantation (SCT) recipients are enrolled. Patients then accrue to cohort 2 based on documented cytomegalovirus (CMV) infection and preemptive treatment with ganciclovir within 90 days after SCT (patients previously accrued to cohort 1 can be accrued to cohort 2 if they develop CMV infection).

* Cohort 1: Patients undergo blood sample collection on approximately days 40, 90, 120, 150, 180, and 360 post transplantation. Samples are analyzed (to determine the development of CMV immunity) for prevalence of CMV-specific cytotoxic T-lymphocytes (CTL) by HLA-peptide tetramer-binding assay (TBA) pp65, with and without in vitro stimulation (IVS). Samples collected on days 40 and 90 are also analyzed by chromium release assay (CRA). Patients suspected of developing CMV viremia may receive ganciclovir according to standard clinical practice.
* Cohort 2: Patients undergo blood sample collection on approximately days 90, 120, 150, 180, and 360 after SCT. Samples are analyzed by TBApp65 staining and for prospective measurement of CMV-specific CTL functions.

All patients undergo routine clinical surveillance for CMV infection on days 21 to 100 after SCT. CMV viral load measurements are obtained twice weekly by CMV-DNA PCR assays on blood cells and plasma and shell-vial blood cultures. In cohort 2, CMV viral load is also determined on days 90 (if not previously as part of cohort 1), 120, 150, 180, and 360. The CMV infection data obtained is then compared with TBA and CTL measurements using HLA-specific tetramers and IVS-induced cytotoxicity assays. Clinical events, such as graft-versus-host disease, underlying disease status, and procedure-related complications are also analyzed and correlated with TBA results.

Stromal cell cultures are obtained from marrow donors at the time of marrow harvest for use as target cells in CTL assays. Donor saliva samples are also obtained for detection of CMV infection by shell-vial method.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria at the City of Hope National Medical Center:

  * Patient who has undergone a matched-related or matched-unrelated allogeneic bone marrow or peripheral blood stem cell transplantation (SCT) for a hematological malignancy (e.g., aplastic anemia or myelodysplastic syndromes)

    * At risk for cytomegalovirus (CMV) infection and disease due to 1 of the following risk factors:

      * CMV-seropositive prior to transplantation
      * Received SCT from a CMV-seropositive donor
  * Donor for matched-related SCT
  * Healthy volunteer evaluated concurrently with SCT recipients to establish normal values for both CMV-seronegative and CMV-seropositive persons
* Any HLA serotypes allowed

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Quantitative determination of HLA-peptide tetramer-binding assay (TBA) pp65 on days 40 and 90 after stem cell transplantation, with and without in vitro stimulation
Comparison of quantitative determination of TBApp65 with concomitant determination of in vitro CMV-specific cytotoxic T-lymphocyte function on days 40 and 90 after stem cell transplantation
Correlation of TBApp65 results with CMV viral loads
Correlation of TBApp65 results with CMV-associated complications

SECONDARY OUTCOMES:
Correlation of TBApp65 results with clinical events, including acute graft-versus-host-disease (GVHD), chronic GVHD, ganciclovir exposure, and survival

CONTACTS AND LOCATIONS:
Overall Officials: John A. Zaia, MD, Principal Investigator — City of Hope Comprehensive Cancer Center

REFERENCES:
- [Derived] Lacey SF, La Rosa C, Kaltcheva T, Srivastava T, Seidel A, Zhou W, Rawal R, Hagen K, Krishnan A, Longmate J, Andersson HA, St John L, Bhatia R, Pullarkat V, Forman SJ, Cooper LJ, Molldrem J, Diamond DJ. Characterization of immunologic properties of a second HLA-A2 epitope from a granule protease in CML patients and HLA-A2 transgenic mice. Blood. 2011 Aug 25;118(8):2159-69. doi: 10.1182/blood-2011-04-349951. Epub 2011 Jun 30. PMID 21719601